CLINICAL TRIAL: NCT03628456
Title: Effect of High Frequency Chest Wall Oscillation Vests on Spirometry Measurements, Comparative Study
Brief Title: Effect of HFCWO Vests on Spirometry Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Biophysics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-01
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Results first posted 2019-11-13 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Cystic Fibrosis; Bronchiectasis
MeSH Terms: conditions — Cystic Fibrosis; Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- AffloVest Monarch Arm (Experimental): Devices placed on highest intensity / highest frequency
  Interventions: Device: International Biophysics AffloVest; Device: Hill-Rom Monarch

INTERVENTIONS:
Device: International Biophysics AffloVest — High-frequency chest wall oscillation vest
Device: Hill-Rom Monarch — High-frequency chest wall oscillation vest

SUMMARY:
The impact of high-frequency chest wall oscillation therapy on spirometry values (Forced Expiratory Volume, Forced Vital Capacity, Peak Expiratory Flow, Forced Expiratory Flow and Tidal Volume is investigated during use of several products and comparing to baseline values

DETAILED DESCRIPTION:
The study will be broken into one (1) arm:

• AffloVest® & Monarch™

Within the arm, the order of products will be randomized.

Baseline spirometry (Forced Expiratory Volume (FEV1), Forced Vital Capacity (FVC), Peak Expiratory Flow (PEF), Forced Expiratory Flow (FEF25-75%) and Tidal Volume (TV)) will be taken at the beginning, middle and end of each series of measurements with each subject, without any device on the subject. A product (AffloVest or Monarch) will be placed onto subject and turned ON to the highest frequency and intensity settings. Then the subject will be given a certain period of time to adjust and spirometry measurements will then be repeated, then the product will be removed and the subject will be allowed a recovery period, then the other product will be placed on the subject, turned ON and spirometry measurements will repeated.

ELIGIBILITY:
Inclusion Criteria:

- Healthy subject, ages 18 - 50

Exclusion Criteria:

* Non-ambulatory
* diagnosed neuromuscular disorder
* currently using any type of oscillation vest therapy
* diagnosed co-morbid condition (i.e. lung cancer, other lung disorder or disease)
* currently enrolled in a medical research study
* non-English speaking
* presence of the following active implantable devices: pacemakers, neurostimulators, infusion pumps, circulatory support devices, implantable cardioverter defibrillators (ICD's), cochlear implants
* presence of head and/or neck injury that has not yet been stabilized
* presence of active hemorrhage with hemodynamic instability

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2019-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W O'Brien, MD, Principal Investigator — PDS Research
Locations (1):
- PDS Research, Kissimmee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AffloVest Monarch Arm
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AffloVest Monarch Arm
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Tidal Volume (TV) Assessed in Participants at Baseline and With Both Devices
Description: Tidal Volume is the normal volume of air displaced between normal inhalation and exhalation, measured using standard sprirometry techniques
Time Frame: 30 minutes
Measure: Mean (Full Range); unit: L
Groups:
- Baseline: Patient baseline result
- AffloVest Arm: AffloVest placed on subject at highest intensity for five (5) minutes
- Monarch Arm: Monarch placed on subject at highest intensity for five (5) minutes
Arm/Group | Baseline | AffloVest Arm | Monarch Arm
Number analyzed (Participants) | 10 | 10 | 10
L | 0.79 [0.36 to 1.87] | 0.93 [0.34 to 2.47] | 1.12 [0.38 to 2.24]

2. Primary Outcome: Peak Expiratory Flow (PEF) Assessed in Participants at Baseline and With Both Devices
Description: Peak Expiratory Flow (PEF) measures the peak flow during a forced exhalation, measured using standard spirometry techniques
Time Frame: 30 minutes
Measure: Mean (Full Range); unit: L/s
Arm/Group | Baseline | AffloVest Arm | Monarch Arm
Number analyzed (Participants) | 10 | 10 | 10
L/s | 7.08 [4.39 to 10.62] | 7.09 [4.38 to 10.32] | 7.68 [4.85 to 11.16]

3. Primary Outcome: Forced Vital Capacity (FVC) Assessed in Participants at Baseline and With Both Devices
Description: Forced Vital Capacity (FVC) is the total amount of air exhaled during the FEV test, measured using standard spirometry techniques
Time Frame: 30 minutes
Measure: Mean (Full Range); unit: L
Arm/Group | Baseline | AffloVest Arm | Monarch Arm
Number analyzed (Participants) | 10 | 10 | 10
L | 3.82 [2.61 to 5.45] | 3.70 [2.48 to 5.45] | 3.83 [2.77 to 5.04]

4. Primary Outcome: Forced Expiratory Volume (1 Second) Assessed in Participants at Baseline and With Both Devices
Description: Forced Expiratory Volume in 1 second (FEV1) measures how much air a person can exhale during a forced breath during the first one (1) second, measured using standard spirometry techniques
Time Frame: 30 minutes
Measure: Mean (Full Range); unit: L
Arm/Group | Baseline | AffloVest Arm | Monarch Arm
Number analyzed (Participants) | 10 | 10 | 10
L | 3.18 [2.15 to 4.73] | 3.04 [2.03 to 4.66] | 3.09 [2.23 to 4.33]

5. Primary Outcome: Forced Expiratory Flow (FEF25-75%) Assessed in Participants at Baseline and With Both Devices
Description: Forced Expiratory Flow (25-75%) is the average flow from the point at which 25% of the FVC has been exhaled to the point at which 75% of the FVC has been exhaled, measured using standard spirometry techniques
Time Frame: 30 minutes
Measure: Mean (Full Range); unit: L/s
Arm/Group | Baseline | AffloVest Arm | Monarch Arm
Number analyzed (Participants) | 10 | 10 | 10
L/s | 3.37 [2.24 to 5.06] | 3.08 [1.85 to 4.90] | 3.05 [2.24 to 4.54]

ADVERSE EVENTS:
Time Frame: 2 hours
Groups:
- AffloVest Arm: AffloVest placed on highest intensity
- Monarch Arm: Monarch placed on highest intensity
Arm/Group | Baseline | AffloVest Arm | Monarch Arm
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/56/NCT03628456/Prot_SAP_000.pdf